CLINICAL TRIAL: NCT03484520
Title: Phase 1b Study of Venetoclax and Dinaciclib (MK7965) in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: A Study of Venetoclax and Dinaciclib (MK7965) in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-183; 2017-003213-26 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2018-03-26; First posted 2018-03-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Cancer - Acute Myeloid Leukemia
Keywords: Cancer, Acute Myeloid Leukemia (AML), venetoclax, dinaciclib, Relapsed/refractory AML, Pharmacokinetics, Venetoclax, Dinaciclib
MeSH Terms: conditions — Neoplasms; Leukemia, Myeloid, Acute; Recurrence | interventions — venetoclax; dinaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax + Dinaciclib (Experimental): Venetoclax and dinaciclib will be administered in combination. Different combinations of dose levels for venetoclax and dinaciclib will be explored.
  Interventions: Drug: Venetoclax; Drug: Dinaciclib

INTERVENTIONS:
Drug: Venetoclax — tablet, oral
  Other Names: ABT-199; GDC-0199
Drug: Dinaciclib — intravenous
  Other Names: MK-7965; SCH-727965

SUMMARY:
An open-label, dose-escalation study to assess safety, pharmacokinetics and efficacy as well as determine the recommended Phase 2 doses of co-administered therapy of dinaciclib and venetoclax for patients with relapsed or refractory Acute Myeloid Leukemia (R/R AML).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) by World Health Organization criteria excluding acute promyelocytic leukemia (APL)-M3.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Participant must have adequate hematologic, renal, and liver function laboratory values as described in the protocol.

Exclusion Criteria:

* Known central nervous system leukemia
* Severe chronic obstructive pulmonary disease (COPD) with hypoxemia
* History of any malignancy within the last 6 months except for those specified in this protocol and low-grade malignancies not requiring active treatment.
* Prior allogeneic stem cell transplant within 6 months of study drug administration and no requirement for graft versus host therapy.
* History of clinically significant medical condition that, in the opinion of the investigator, would adversely affect participation in this study.
* Known active infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* History of tumor lysis syndrome (TLS) due to previous exposure to venetoclax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Tmax of Venetoclax | Approximately 29 days after first dose of study drug
  Time to maximum plasma concentration (Tmax) of venetoclax.
Recommended Phase 2 Dose (RPTD) of co-administered Dinaciclib and Venetoclax | Minimum first cycle of dosing (21 days)
  Tthe RPTD of co-administered venetoclax and dinaciclib will be determined during the dose escalation phase of the study. RPTD will be determined using available safety and pharmacokinetics data.
Cmax of Venetoclax | Approximately 29 days after first dose of study drug
  Maximum observed plasma concentration (Cmax) for Venetoclax.
AUCt of Venetoclax | Approximately 29 days after first dose of study drug
  Area Under the Plasma Concentration-time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUCt)
AUC0-24 Post-dose of Venetoclax | Approximately 29 days after first dose of study drug
  Area under the plasma concentration-time curve from 0 to 24 hours (AUC24) post-dose of venetoclax.
Cmax of Dinaciclib | Approximately 29 days after first dose of study drug
  Maximum plasma concentration (Cmax) of dinaciclib.
Half-life (t1/2) of Dinaciclib | Approximately 29 days after first dose of study drug
  Half-life (t1/2) of dinaciclib.
AUCt Post-dose of Dinaciclib | Approximately 29 days after first dose of study drug
  Area under the plasma concentration-time curve from time zero to time t (AUCt) post-dose dinaciclib.
AUC0-∞ of Dinaciclib | Approximately 29 days after first dose of study drug
  Area under the plasma concentration-time curve from 0 to infinity (AUC0-∞) post-dose of dinaciclib.
Clearance of Dinaciclib | Approximately 29 days after first dose of study drug
  Clearance (CL) of dinaciclib.

SECONDARY OUTCOMES:
Complete Response (CR) Rate | Up to approximately 18 months
  CR is defined as the proportion of participants with documented complete response (CR) based on International Working Group (IWG) criteria.
Composite CR Rate (CR + CRi) | Up to approximately 18 months
  Composite is defined as CR + CRi (CR with incomplete blood count recovery) based on IWG criteria.
Objective Response Rate (ORR) | Up to approximately 18 months
  ORR is defined as the proportion of participants with documented partial response (PR) or better (CR + CRi + partial response [PR]) based on IWG criteria.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- United States (7):
  - University of Arkansas /ID# 200016, Little Rock, Arkansas
  - David Geffen School of Medicin /ID# 200015, Los Angeles, California
  - The University ofChicago /ID# 200017, Chicago, Illinois
  - University of Maryland School of Medicine /ID# 204015, Baltimore, Maryland
  - Wake Forest Baptist Medical Center /ID# 200288, Winston-Salem, North Carolina
  - The Ohio State University /ID# 200668, Columbus, Ohio
  - University of Texas MD Anderson Cancer Center /ID# 205215, Houston, Texas
- Australia (3):
  - Gold coast University Hospital /ID# 202759, Southport, Queensland
  - Royal Hobart Hospital /ID# 202763, Hobart, Tasmania
  - Monash Medical Centre /ID# 202762, Melbourne, Victoria
- Spain (3):
  - Hospital Universitario Ramon y Cajal /ID# 201729, Madrid
  - Hospital Universitario de Salamanca /ID# 201728, Salamanca
  - Hospital Universitario y Politecnico La Fe /ID# 202318, Valencia

IPD SHARING:
Plan to Share IPD: No